CLINICAL TRIAL: NCT04433325
Title: COVID-19 Critically Ill Patients' Evolution After Medical Transport by Train From Paris Intensive Care Units to West of France Intensive Care Units
Acronym: TOCCIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_3091_TOCCIP
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Intensive Care Unit Syndrome
Keywords: Medical transport by train
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients transferred: Patients transferred from Paris's Intensive Care Units
- Patients not transferred: Patients admitted in Intensive Care Units with no transfer from Paris

SUMMARY:
Since early 2020, France knows a sanitary crisis with a massive influx of COVID-19 patients admitted in Intensive Care Units (ICU). It led to a saturation of the French health system, especially in some geographic areas such as East of France or Paris region. Therefore, authorities decided to transfer some critically ill patients from these crowded ICUs to less busy regional ICUs. it was done for the first time by medical train transportation. Knowing that the investigators lack experience regarding this type of medical evacuation, regarding the high number of transferred patients, with such a logistic effort, the investigators decided to study this phase of the COVID-19 sanitary crisis in order to draw a feedback. So far, there are no data in the literature regarding this topic.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* COVID-19 positive patients admitted in Intensive Care Unit between 15/03/2020 and 15/04/2020
* Patients (or legal representative) with no opposition to inclusion in medical research protocol
* Regarding case group : Patients transferred from Paris's ICU
* Regarding case control group : Patients admitted in ICU with no transfer from Paris

Exclusion Criteria:

- > 18 years under legal protection and patients with liberty restriction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients admitted in Intensive Care Unit between 15/03/2020 and 15/04/2020
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
number of death | at Intensive Care Units discharge, an average of 1 months
  to evaluate mortality

SECONDARY OUTCOMES:
number of infections | from date of admission until Intensive Care Units discharge, assessed up to 1 months
  to evaluate morbidity
number of days of mechanical ventilation | from date of admission until Intensive Care Units discharge, assessed up to 1 months
number of days of sedation | from date of admission until Intensive Care Units discharge, assessed up to 1 months
number of days of use of neuromuscular blocking agents | from date of admission until Intensive Care Units discharge, assessed up to 1 months
number of days of vasopressor use | from date of admission until Intensive Care Units discharge, assessed up to 1 months
number of days in Intensive Care Units | from date of admission until Intensive Care Units discharge, assessed up to 1 months
number of days in hospital | from date of admission until hospital discharge, assessed up to 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Painvin, Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - CHU Poitiers, Poitiers
  - CHU Tours, Tours